CLINICAL TRIAL: NCT07256132
Title: The Efficacy of Erector Spinae Plane Block for the Relief of Chronic Pain in Cases of Degenerative Disc Diseases.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0305626
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain in Degenerative Disc Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injected patients (Experimental)
  Interventions: Procedure: erector spinae plane block
- care provider (No Intervention)

INTERVENTIONS:
Procedure: erector spinae plane block — erector spinae plane block
  Arms: injected patients

SUMMARY:
Erector Spinae Plane Block is an effective pain therapy technique to relieve chronic low back pain in cases of degenerative disc disorders.

DETAILED DESCRIPTION:
This study will be conducted on 40 adult patients with degenerative disc disease (DDD) of the lumbar spine and admitted to the Neurosurgery Department at Alexandria Main University Hospital aged between 30 and 65 years old with Visual analog scale more than or equal to 4 not responding to conservative treatment, patients having grade 0, 1 or 2 lumbar disc degeneration without disc bulge or prolapse by X-ray and MRI with loss or decreased lumbar lordosis, patients with black disc and contained disc bulge on magnetic resonance imaging (MRI) and patients with grade I degenerative spondylolisthesis provided that the canal dimensions are normal or with mild stenosis. Patients with severe sciatic pain, patients with more than two levels of DDD of the lumbar region or with isthmic spondylolisthesis and high-grade instability, or patients with disc fragments encroaching upon the exit foramina and nerve root or with severe canal stenosis, also those with central obesity, recurrent disc prolapse or with previous abdominal surgery were excluded from the study. Steroid injection will avoided in patients with immunosuppression or uncontrolled diabetes.

Both a full history taking and a clinical examination will be completed. All patients underwent an MRI of the lumbar region for evaluation. Routine laboratory and other lab investigations will conducted.

ELIGIBILITY:
Inclusion Criteria:

* This study was conducted on 40 adult patients with degenerative disc disease (DDD) of the lumbar spine and admitted to the Neurosurgery Department at Alexandria Main University Hospital aged between 30 and 65 years old with Visual analog scale more than or equal to 4 not responding to conservative treatment, patients having grade 0, 1 or 2 lumbar disc degeneration without disc bulge or prolapse by X-ray and MRI with loss or decreased lumbar lordosis, patients with black disc and contained disc bulge on magnetic resonance imaging (MRI) and patients with grade I degenerative spondylolisthesis provided that the canal dimensions are normal or with mild stenosis

Exclusion Criteria:

* Patients with severe sciatic pain, patients with more than two levels of DDD of the lumbar region or with isthmic spondylolisthesis and high-grade instability, or patients with disc fragments encroaching upon the exit foramina and nerve root or with severe canal stenosis, also those with central obesity, recurrent disc prolapse or with previous abdominal surgery were excluded from the study. Steroid injection was avoided in patients with immunosuppression or uncontrolled diabetes.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 8 weeks
  otal scores range from 0 to 10 (based on a scale of 0 to 2 for five items), with a higher score indicating more severe pain.

SECONDARY OUTCOMES:
Oswestry disability index | 8 weeks
  a condition-specific functional measure used to assess the symptoms and severity of low back pain disablement and its impact on patient functional activities

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided